CLINICAL TRIAL: NCT04396327
Title: A Randomized, Double-Blind, Single-Dose, 2-Way Cross-Over Study to Assess the Pharmacodynamic Effects of SM-1 vs. Active Comparator in a 3-Hour Phase Advance Model of Transient Insomnia
Brief Title: SM-1 vs. an Active Comparator in A Model of Transient Insomnia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sequential Medicine Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SM-A-07
Record Dates: First submitted 2020-05-08; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-04

CONDITIONS: Transient Insomnia
Keywords: Short term Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study will be double-blind. Neither study subjects nor study personnel will have knowledge of the treatments administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Comparator: 2-Drug Combination (Active Comparator): 50 mg diphenhydramine and 0.5 mg lorazepam
  Interventions: Drug: Active Comparator
- Active Treatment: SM-1 3-Drug Combination (Experimental): 3-drug combination product containing 50 mg diphenhydramine, 5 mg zolpidem and 0.5 mg lorazepam
  Interventions: Drug: SM-1

INTERVENTIONS:
Drug: SM-1 — diphenhydramine, zolpidem and lorazepam
  Arms: Active Treatment: SM-1 3-Drug Combination
Drug: Active Comparator — diphenhydramine and lorazepam
  Arms: Active Comparator: 2-Drug Combination

SUMMARY:
The purpose of this study is to investigate the effectiveness, safety and tolerability of a combination drug product (SM-1) containing diphenhydramine, zolpidem and lorazepam, in adult participants who sometimes have difficulty in falling asleep or staying asleep, but who do not have chronic insomnia. Participants will receive SM-1 or a combination of diphenhydramine and lorazepam during 2 one-night stays at a sleep center.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of a combination drug product containing 50 mg diphenhydramine, 5 mg zolpidem and 0.5 mg lorazepam on total sleep time, and to determine the contribution of zolpidem to the combination, using a 3-hour Phase Advance model of sleep challenge with 8 hours of polysomnographic (PSG) recording. This is a 2-arm, 2-period crossover trial including the 3-drug investigational product and a 2-drug comparator. The 2 arms are: investigational combination product, and a 2-drug comparator containing diphenhydramine and lorazepam but not zolpidem. Participants will be adults who sometimes have difficulty falling asleep or staying asleep, but who are generally healthy and do not have chronic insomnia or sleep apnea.

A total of 14 subjects are planned to enroll in the study. Subjects who qualify for participation will be asked to keep a sleep diary to document their sleep times leading up to their first overnight stay in the sleep center and during the study. Subjects will be asked to spend at least 7.5 hours in bed at a regular bedtime during the study. Qualifying participants also will not anticipate traveling across 3 time zones, be involved in night shift work, or significant disruptions in their sleep schedules during the study. The study requires 2 one-night stays in a sleep center in New York City, for administration of the study treatments and PSG & EEG measurements. Qualifying subjects will anticipate being able to return to the sleep center, located in Manhattan, for a total of 3 visits, including initial screening and 2 treatment times.

Subjects will receive a follow up phone call from study staff 3 days after final dose of study medication.

During each sleep center visit, subjects will arrive to the sleep center approximately 5 hours prior to their average usual bedtime and will be given their study treatment. Their sleep will be monitored for 8 hours. Each subject will receive both treatments, although the sequence of the 2 treatments will be randomized. Both subjects and study personnel monitoring the subjects will be blinded to the identity of the treatment administered at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25 and 55 years
2. Body mass index (BMI) between 19 and 32 kg/m2
3. Report previous history of occasional difficulty falling asleep or staying asleep, but not currently having difficulty sleeping;
4. Regular, habitual bedtime between 21:00 and 24:00, routinely spend at least 7.5 and no more than 9.0 hours in bed nightly and a bedtime that does not vary by more than 2 hours over the course of the week.
5. Good general health
6. Females of childbearing potential must be using an acceptable method of contraception, have a negative serum pregnancy test at screening and have a negative urine pregnancy test before randomization and prior to each Treatment Period.
7. Female subjects who have been surgically sterilized are eligible if they have a negative serum pregnancy test at screening and negative urine pregnancy test at check-in or are post-menopausal or have had a complete hysterectomy;
8. Male subjects must use an acceptable method of contraception during the course of the study and for the 90 days following the last dose of study medication.
9. Obtain signed informed consent
10. Able to stay in the clinical research unit for 1 overnight stay during each treatment period
11. No alcohol on check-in days
12. Refrain from the use of alcohol and from napping on site check-in days
13. A recent history of napping of no more than once per week.

Exclusion Criteria:

1. Clinically significant, acute illness within 14 days prior to screening
2. Clinically significant, unstable medical illness;
3. Evidence or history of clinically significant allergic hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic or neurological disease;
4. History of cancer or diabetes;
5. A sitting blood pressure > 140/90 millimeters mercury (mm/Hg) at screening;
6. Heart rate > 100 beats per minute (BPM) at screening;
7. Clinically significant psychiatric illness, including chronic psychiatric illness or the history or presence of any Axis I condition;
8. Subject has homicidal ideation/intent, per the investigator's clinical judgment, or has suicidal ideation with some intent to act within 6 months prior to the start of the screening phase, per the investigator's clinical judgment or based on the C-SSRS
9. History or presence of chronic pain;
10. Lifetime history of seizure disorder or serious head injury;
11. Clinically significant sleep disorder, including chronic insomnia, sleep apnea, narcolepsy, parasomnia, restless leg syndrome or circadian rhythm disorder;
12. Slept in a sleep laboratory at any time prior to Screening.
13. STOP-BANG sleep apnea questionnaire >/= to 3 at Screening;
14. Epworth Sleepiness Scale (ESS) score >10 at screening;
15. Any condition that may affect drug absorption;
16. Travel across more than three time zones or shift worker
17. Any clinically significant abnormal finding on physical examination, vital signs or clinical laboratory tests,
18. History of allergies, or known sensitivity, hypersensitivity, or adverse reaction to any drug similar to diphenhydramine, zolpidem or lorazepam;
19. Pregnant or lactating females;
20. Positive serum or urine pregnancy test
21. Positive urine drug screen
22. Recent history or current evidence of alcohol or drug abuse
23. Regular consumption of "large amounts" of xanthine-containing substances (i.e., [equivalent to approximately 2 - 3 cups of regular coffee] or equivalent amounts of xanthine-containing substances);
24. Usual consumption of more than 14 units of alcohol per week.
25. Use of more than 10 cigarettes or equivalent per day of any product containing nicotine or routinely smokes during sleep period.
26. Stopped smoking or in a smoking cessation program within 90 days of screening;
27. Use of restricted concomitant medications, any prescription drug, OTC medication, grapefruit, grapefruit juice, herbal preparation or food supplement, excluding vitamins, acetaminophen or hormonal contraceptives

29. Exposure to any investigational drug or to diphenhydramine, zolpidem or lorazepam or other drugs of the same pharmaceutical classes within 30 days of screening 30. Positive alcohol or drug test

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2020-05-27 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Latency to Persistent Sleep (LPS) | 8 hours
  Time it takes to fall asleep

SECONDARY OUTCOMES:
Wakefulness | 8 hours
  Time spent awake in minutes
Subjective Sleep Latency | 8 hours
  Time it takes to fall asleep in minutes
Adverse Events | 8 hours
  Safety and tolerability assessed in terms of the incidence of AEs

OTHER OUTCOMES:
Total Sleep Time (TST) | 8 hours
  Duration of sleep in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Maha Ahmad, MD, MMSc, Principal Investigator — Clinilabs Drug Development Corporation
Locations (1):
- Clinilabs Drug Development Corporation, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No